Official Title: Evaluation of PEEK Versus Titanium Bar Attachments with Implant-Assisted Mandibular Complete Overdenture Fabricated by CAD/CAM Technology NCT Number: Not yet assigned Document Date: February 20, 2024

### **Clinical Trial Protocol**

Study Type: Interventional (Clinical Trial)

# **Study Design:**

• Allocation: Randomized

• Intervention Model: Parallel Assignment

• Masking: None (Open Label)

• Primary Purpose: Treatment

## **Study Population:**

• Total Sample Size: 12 patients

• Age Range: 40–60 years

### • Inclusion Criteria:

- o Completely edentulous mandibular arch
- o Adequate bone quantity and quality for implant placement
- o Class I maxilla-mandibular relationship
- Sufficient inter-arch space (≥25 mm)
- Good oral hygiene

## • Exclusion Criteria:

- Systemic diseases affecting tissue healing
- History of radiation therapy in head/neck region
- Neurological or psychological disorders affecting oral hygiene
- Parafunctional habits
- Heavy smoking, alcoholism, or drug abuse

### **Study Groups / Interventions:**

- **Group I (Control):** CAD/CAM Titanium bar attachment mandibular overdenture (6 patients)
- **Group II (Study):** CAD/CAM PEEK bar attachment mandibular overdenture (6 patients)

#### **Outcome Measures:**

### • Primary Outcome:

• Retention force of mandibular overdenture measured in Newtons using a digital force meter at insertion, 6 months, and 1 year

## • Secondary Outcomes:

- Marginal bone loss around implants measured via digital periapical X-rays at insertion, 6 months, and 1 year
- Bar deviation assessed digitally by STL file superimposition at 6 months and 1 year

## **Study Setting:**

Prosthodontics Department, Faculty of Dentistry, Tanta University, and CAD/CAM laboratory

### **Ethical Consideration:**

• Informed consent will be obtained from all participants according to the guidelines of the Research Ethics Committee, Faculty of Dentistry, Tanta University